CLINICAL TRIAL: NCT07213752
Title: Diode Laser-Assisted Periodontal Therapy Enhances Clinical Outcomes for Deep Periodontal Pockets in Smokers: A Randomized Clinical Trial
Brief Title: Diode Laser-Assisted Periodontal Therapy Enhances Clinical Outcomes for Deep Periodontal Pockets in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Deniz irem Atasoy Erdogan, Deniz Irem Atasoy Erdoğan, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-DIAE-01
Record Dates: First submitted 2025-09-29; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis; Periodontitis Stage III; Periodontal Disease; Diode Laser Therapy; Smoking; Malondialdehyde
Keywords: adjunctive periodontal treatment; diode laser therapy; non-surgical periodontal therapy; smokers with periodontitis; malondialdehyde; 8-hydroxy-2'-deoxyguanosine
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Smoking | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To ensure allocation concealment and maintain the masked design, the following protocol was applied: After diagnosis at the Department of Oral Diagnosis and Radiology, baseline periodontal records and anamnesis were documented, and each patient was assigned a unique ID. Eligible participants underwent baseline clinical measurements (D.İ.A) and saliva sampling. Patients were then randomly allocated to SRP (n=17) or SRP+DL (n=16) using a computer-generated program (Sealed Envelope Ltd.) by an independent clinician not involved in the study. One week later, SRP and diode laser procedures were performed by the same clinician (D.İ.A). For blinding, all clinical files were anonymized and coded by the study supervisor (S.S.H). Statistical analyses were conducted by a blinded statistician without access to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stage III Grade C :Non surgical periodontal therapy and an adjunct diode laser use (Experimental)
  Interventions: Device: Diode Laser Application in Deep Periodontal Pockets; Procedure: Professional Mechanical Plaque Removal; Procedure: Scaling and Root Planing
- Stage III Grade C :Non surgical periodontal therapy (Experimental)
  Interventions: Procedure: Professional Mechanical Plaque Removal; Procedure: Scaling and Root Planing

INTERVENTIONS:
Device: Diode Laser Application in Deep Periodontal Pockets — A 940 nm indium-gallium-aluminum-phosphate diode laser (Ezlase, Biolase, USA) with a 400 μm fiber was used in contact mode at 1.5 W, pulse 20/20 ms, 20 s/cm², power density 1.061 W/cm², and 15 J/cm² energy in deep periodontal pockets.
  Arms: Stage III Grade C :Non surgical periodontal therapy and an adjunct diode laser use
Procedure: Professional Mechanical Plaque Removal — Professional mechanical removal of supragingival plaque and calculus
Procedure: Scaling and Root Planing — Subgingival scaling and root planing

SUMMARY:
This study investigated the adjunctive effects of diode laser therapy in smokers with severe periodontitis. Thirty-three patients were randomized to non-surgical periodontal therapy (SRP) with or without diode laser. Clinical parameters and salivary oxidative stress markers (MDA, 8-OHdG) were assessed at baseline, 1, and 3 months. Both groups showed improvements, but SRP+DL resulted in significantly greater reductions in deep pockets, PISA, PESA, PI, and MDA at 3 months. These findings suggest that diode laser therapy may enhance conventional treatment by improving clinical outcomes and reducing oxidative stress in smokers with severe periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* no periodontal treatment within the previous 6 months;
* no use of antibiotics within the previous 3 months;
* no systemic disease and alcohol drinkers, or drug users;
* no use of anti-inflammatory drugs within the past 3 months;
* no pregnancy;
* no use of hormonal contraceptives; and
* current smokers with a history of smoking ≥10 cigarettes per day for at least one year.

Exclusion Criteria:

* Patients with <20 teeth, grade III tooth mobility, partial dentures, or fixed prostheses were excluded. Additionally, those with dental implants or peri-implant diseases were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Dept (PPD) | Through study completion, an average of 3 months.
  The probing pocket dept was assessed on six tooth surfaces, inluding the mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual areas of each tooth.
Periodontal Epithelial Surface Area (PESA) | Through study completion, an average of 3 months.
  PESA represents the total epithelial surface area in periodontal pockets.
Periodontal Inflamed Surface Area (PISA) | Through study completion, an average of 3 months.
  PISA quantifies the inflamed portion of this surface area by integrating only sites exhibiting BOP, both measured in mm2.
Salivary Malondialdehyde Levels | Through study completion, an average of 3 months.
  Evaluation of salivary malondialdehyde levels.
Salivary 8-hydroxy-2'-deoxyguanosine Levels | Through study completion, an average of 3 months.
  Evaluation of salivary 8-hydroxy-2'-deoxyguanosine levels.
PPD ≥4 mm, site-specific PPD (ssPPD) | Through study completion, an average of 3 months.
  For sites with PPD ≥4 mm, site-specific PPD (ssPPD) values was calculated.
PPD ≥4 mm, site spesific CAL (ssCAL) | Through study completion, an average of 3 months.
  For sites with PPD ≥4 mm, site spesific CAL (ssCAL) values were also calculated.
PPD ≥4 mm, site-specific PISA (ssPISA) | Through study completion, an average of 3 months.
  For sites with PPD ≥4 mm, site-specific PISA (ssPISA) values were calculated.
PPD ≥4 mm, site-specific PESA (ssPESA) | Through study completion, an average of 3 months.
  For sites with PPD ≥4 mm, site-specific PESA (ssPESA) values were calculated.

SECONDARY OUTCOMES:
Plaque Index (PI) | Through study completion, an average of 3 months.
  The plaque index was assessed on six tooth surfaces, inluding the mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual areas of each tooth.
Bleeding on Probing (BOP) | Through study completion, an average of 3 months.
  The bleeding on probing index was assessed on six tooth surfaces, inluding the mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual areas of each tooth.
Clinical Attachment Level (CAL) | Through study completion, an average of 3 months.
  The clinical attachment level was assessed on six tooth surfaces, inluding the mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual areas of each tooth.
Gingival Index (GI) | Through study completion, an average of 3 months.
  The gingival index was assessed on six tooth surfaces, inluding the mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual areas of each tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Dentistry Department of Periodontology, Konya, Selçuklu, Turkey (Türkiye)